CLINICAL TRIAL: NCT02556242
Title: From Malaria Control to Sustainable Elimination: Cluster Randomised Trial Comparing Targeted Versus Generalised Vector Control in South Africa
Brief Title: Targeted Indoor Residual Spraying Against Malaria
Acronym: TIRS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Witwatersrand, South Africa (Other); National Department of Health, South Africa (Unknown); Medical Research Council (Other Government); National Institute for Communicable Diseases, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPIDZC8610
Record Dates: First submitted 2015-09-07; First posted 2015-09-22 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Malaria
Keywords: vector control; insecticide
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targeted indoor residual spraying (Experimental): The intervention arm of the trial will receive Indoor Residual Spraying delivery through targeted spraying in the neighbourhood of recent local cases only.
  Interventions: Other: Targeted indoor residual spraying
- Generalised Indoor residual spraying (Active Comparator): The reference (control) arm of the trial will receive Indoor Residual Spraying through generalised annual spraying of all structures, as is the current standard practice.
  Interventions: Other: Generalised Indoor residual spraying

INTERVENTIONS:
Other: Targeted indoor residual spraying — IRS is carried out in neighbourhoods of cases
  Arms: Targeted indoor residual spraying
Other: Generalised Indoor residual spraying — IRS is carried out as normally practiced
  Arms: Generalised Indoor residual spraying

SUMMARY:
Since 2000, annual numbers of malaria cases in South Africa have sharply declined to about 5,000, with case numbers fairly stable since 2007. The principal malaria prevention strategy has consisted of generalised Indoor Residual Spraying (IRS) of all houses in malaria endemic districts. As recent case data indicate that the levels of transmission in many districts have been reduced to very low levels, the continuation of untargeted IRS in areas where there is little or no evidence of recent transmission may be unwarranted. Efforts to eliminate malaria will only be sustainable if mass prevention efforts can be scaled down in an evidence-based manner, whilst maintaining or enhancing high sensitivity of the surveillance system of the disease. This trial will provide scientific evidence for targeted malaria prevention responding to localised transmission in pre-elimination settings, compared to continuation of generalised IRS of all houses.

Two methods of IRS delivery for community malaria prevention will be compared through an open-label cluster-randomised trial consisting of two study arms with 30 clusters per arm of approximately 8,000 inhabitants per cluster.

Comparison is on the basis of non-inferiority by showing that malaria incidence in the targeted IRS arm is no higher than malaria incidence in the generalised IRS arm within a specified margin of difference, and on the basis of superiority showing that the proportion of houses targeted for spraying is higher in the intervention than the reference arm. Neighbourhood investigation in response to each locally acquired case in the intervention arm, and comparison neighbourhoods in the reference arm, will include testing for antibody sero-conversion to malarial antigens to assess whether cases arise in communities with long term exposure to malaria parasites.

The trial will be carried out in the South African provinces of Limpopo and Mpumalanga, in localities which have average reported incidence of malaria of <5 cases per 1000 per annum over the past five years.

DETAILED DESCRIPTION:
Two methods of IRS delivery for malaria prevention, targeted spraying versus annual generalised spraying, will be compared through an open-label cluster randomised trial consisting of two trial arms with 30 clusters per arm. Clusters will be artificial constructs made up of groups of spray localities or complete wards to comprise populations of about 5,000 to 10,000 persons. The unit of randomisation will be the cluster.

The intervention arm of the trial will receive IRS delivery through targeted reactive spraying in the neighbourhood of recent local cases only; the reference (control) arm of the trial will receive IRS through generalised annual spraying of all structures as per standard current practice.

Comparison will be on the basis of non-inferiority by showing that malaria incidence in the targeted IRS arm is no higher than malaria incidence in the generalised IRS arm within a specified margin of difference, and on the basis of superiority showing that the proportion of houses sprayed, of those targeted for spraying, is higher in the intervention than the reference arm. Neighbourhood investigation in response to each locally acquired case in the intervention arm, and comparison neighbourhoods in the reference arm will include testing for antibody sero-conversion to malarial antigens to assess whether cases arise in communities with long term exposure to malarial parasites.

ELIGIBILITY:
Inclusion criteria

1. Entire communities of approximately 8000 persons
2. Residents in malaria endemic districts of Limpopo and Mpumalanga Province
3. Areas with local malaria incidence <5 cases per 1000 per year on average over 5 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 393387 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Malaria incidence, by routine passive case detection, of clinical malaria (fever ≥37.5°C, or history of fever (48 hours), in the presence of parasitaemia confirmed by RDT or microscopy). | Communities will be followed for up to 20 months

SECONDARY OUTCOMES:
Intervention costs per 1,000 households and cost-effectiveness of reactive, targeted indoor residual spraying (TIRS) compared to generalised IRS (GIRS) | Up to 20 months
  Cost of spray operations will be determined in each study arm
Proportion of structures targeted for IRS unsprayed | Up to 20 months whenever reactive spraying is triggered
Household compliance (not painting, washing, re-plastering ) | By cross sectional household survey after 18 months
  In a representative sample household survey in all clusters, a questionnaire will be used in which householders will be asked whether they painted, re-plastered or washed walls after spraying
Householder acceptability of IRS | By cross sectional household survey after 18 months
  In a representative sample household survey in all clusters, a questionnaire will be used in which householders will be asked whether they want their house sprayed with insecticide in future
If unsprayed, proportions due to refusals, spray teams not making contact and spray teams not calling back | By cross sectional household survey after 18 months
  In a representative sample household survey in all clusters, a questionnaire will be used in which householders whose houses remained unsprayed will be asked whether this was because they refused or because spray teams did not make contact or did not call back if they were away
Sero-prevalence of antibodies to malaria antigens AMA-1 and MSP-1-19 | By cross sectional household survey after 18 months
  In a representative sample household survey in all clusters, a filter paper dried blood spot a will be taken from a sample of individuals of all ages, subject to informed written consent

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Coetzee, Phd, Principal Investigator — University of Witwatersrand, South Africa; Immo Kleinschmidt, Phd, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- South Africa (2):
  - Provincial Malaria Control Programme, Tzaneen, Limpopo
  - Provincial Malaria Control Programme, Mbombela, Mpumalnga

REFERENCES:
- [Derived] Bath D, Cook J, Govere J, Mathebula P, Morris N, Hlongwana K, Raman J, Seocharan I, Zitha A, Zitha M, Mabuza A, Mbokazi F, Machaba E, Mabunda E, Jamesboy E, Biggs J, Drakeley C, Moonasar D, Maharaj R, Coetzee M, Pitt C, Kleinschmidt I. Effectiveness and cost-effectiveness of reactive, targeted indoor residual spraying for malaria control in low-transmission settings: a cluster-randomised, non-inferiority trial in South Africa. Lancet. 2021 Feb 27;397(10276):816-827. doi: 10.1016/S0140-6736(21)00251-8. PMID 33640068